CLINICAL TRIAL: NCT02382627
Title: Choroidal Thickness in Optic Neuropathy
Status: Terminated | Type: Observational
Why Stopped: poor enrollment
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 14-2348
Record Dates: First submitted 2015-03-02; First posted 2015-03-09 (Estimated); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Optic Nerve Disorders
MeSH Terms: conditions — Optic Nerve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This study plans to learn more about the thickness of the choroid in patients with optic neuropathy. The choroid is a layer of blood vessels that supplies oxygen and nourishment to the outer layers of the retina. Patients are being asked to be in this research study because they have optic neuropathy and are receiving care at the University of Colorado Hospital.

ELIGIBILITY:
Inclusion criteria:

* age greater than 18 years,
* diagnosis of optic neuropathy,
* willing and able to sign an informed consent.

Exclusion criteria:

* steroid use within the past 4 weeks,
* inability to cooperate with optical coherence tomography (OCT) testing,
* relevant ocular comorbidities in the affected or unaffected eye, such as

  * glaucoma,
  * uveitis,
  * optic nerve hypoplasia,
  * age related macular degeneration,
  * refractive error greater than 5 spherical diopters.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 patients with optic neuropathy seen in the ophthalmology or neuro-ophthalmology clinics at the University of Colorado will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2015-03; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Difference of the subfoveal and parafoveal choroidal thickness in affected and unaffected eye of the same patient. | 1 time

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Bennett, MD, Principal Investigator — 303-724-6450
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States